CLINICAL TRIAL: NCT02219230
Title: Outcomes Associated With Use of Passive, Adaptive, and Active Prosthetic Knees in Persons With Unilateral, Transfemoral Amputation: a Randomized Crossover Trial
Brief Title: Use of Passive, Adaptive, and Active Prosthetic Knees in Persons With Unilateral, Transfemoral Amputation
Acronym: OPK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Össur Iceland ehf (Industry)
Responsible Party: Principal Investigator, Brian Hafner, Associate Professor, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: Single
Other Study IDs: 40660-A; A62089 (Other: University of Washington)
Record Dates: First submitted 2014-07-29; First posted 2014-08-18 (Estimated); Last update posted 2015-12-28 (Estimated); Status verified 2015-12

CONDITIONS: Transfemoral Amputation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Prosthetic knee (Experimental): Subjects crossed over between interventions (three different prosthetic knees). Knee conditions include 1) Active knee (Ossur Power Knee II); 2) Adaptive knee (Ossur Rheo); and 3) Passive knee (Various manufacturers)
  Interventions: Device: Active knee (Ossur Power Knee II); Device: Adaptive knee (Ossur Rheo); Device: Passive knee (Various manufacturers)

INTERVENTIONS:
Device: Active knee (Ossur Power Knee II) — Prosthetic knee with active control system.
  Other Names: Power knee; Motorized knee
Device: Adaptive knee (Ossur Rheo) — Prosthetic knee with adaptive control system.
  Other Names: Magnetorheological knee; Microprocessor knee
Device: Passive knee (Various manufacturers) — Prosthetic knee with mechanical control system.
  Other Names: Mechanical knee; Hydraulic knee; Pneumatic knee

SUMMARY:
The goals of this study are to assess measured, observed, and self-reported outcomes achieved through the use of passive (mechanical), active(motorized) and adaptive (magnetorheological) prosthetic knee control systems in individuals with unilateral, transfemoral amputation.

DETAILED DESCRIPTION:
An interrupted time-series trial with pre/post baseline assessments, randomized crossover of interventions, and within-phase repeated measures is used to evaluate and compare the effectiveness of the Össur Power Knee II and the Össur Rheo Knee in individuals with unilateral, transfemoral amputation. A rigorous and clinically-meaningful experimental protocol is applied to verify study participants receive appropriate training, experience, and assessment in each knee condition. A suite of standardized and ad-hoc physical performance tests, patient-reported questionnaires, and monitoring technologies were carefully selected to assess important, clinically-relevant participant outcomes. Comparative effectiveness of three prosthetic knee interventions are evaluated using direct measurement (i.e., timed tests), observed clinical ratings (i.e., subjective assessments of gait quality) and self-report instruments (i.e., health status surveys). Analyses will focus on identifying differences between control system technologies inherent to each type of prosthetic knee (i.e., passive [mechanical], adaptive [magnetorheological], and active [power]). Outcomes will be used to establish recommendations for which activities and patients knees are most appropriate or likely to produce a desired effect.

ELIGIBILITY:
Inclusion Criteria:

* age 45 - 75
* body weight less than 275lbs
* unilateral amputation between the hip and knee
* amputation due to non-vascular causes
* no other major limb amputations
* amputation occurred at least 2 years prior
* stable limb volume (i.e., at least 6 months on an unmodified prosthetic socket)
* intact skin tissue without open wounds or sores for at least 2 months
* physiologically stable medical condition (i.e., non-degenerative)
* possession and regular (i.e., daily) use of a prosthesis with a prosthetic knee with non-microprocessor (i.e., mechanical or fluid) stance control
* Medicare functional classification level (MFCL or "K-level") 3

Exclusion Criteria:

* expect to receive or are expected to require a replacement prosthetic socket within 15 months
* complete reliance on an assistive device (i.e., cane or walker) for ambulation

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-06; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Timed Up and Go | Change from Baseline (mean score at weeks 1, 2, 3, and 4) to Follow-Up (mean score at weeks 8, 12, 16, 20, 24, and 28)
  Timed performance test that measures rising from a chair, walking 3m, and returning to a seated position.
Timed Ramp Test | Change from Baseline (mean score at weeks 1, 2, 3, and 4) to Follow-Up (mean score at weeks 8, 12, 16, 20, 24, and 28)
  Timed performance test that involves walking up and down a 14ft ramp.
Timed Stair Test | Change from Baseline (mean score at weeks 1, 2, 3, and 4) to Follow-Up (mean score at weeks 8, 12, 16, 20, 24, and 28)
  Timed performance test that involves walking up and down 6 steps.
Step activity | Change from Baseline (mean score at weeks 1, 2, 3, and 4) to Follow-Up (mean score at weeks 8, 12, 16, 20, 24, and 28)
  Average daily step counts measured by an accelerometer-based device.
Obstacle course time | Change from Baseline (mean score at weeks 1, 2, 3, and 4) to Follow-Up (mean score at weeks 8, 12, 16, 20, 24, and 28)
  Time to walk a 1/2-mile outdoor walking course.

SECONDARY OUTCOMES:
Reported Falls | Change from Baseline (mean score at weeks 1, 2, 3, and 4) to Follow-Up (mean score at weeks 8, 12, 16, 20, 24, and 28)
  Self-report phone survey.
Prosthesis Evaluation Questionnaire (PEQ) | Change from Baseline (mean score at weeks 1, 2, 3, and 4) to Follow-Up (mean score at weeks 8, 12, 16, 20, 24, and 28)
  Self-report computerized survey (12 questions)
Activities Specific Balance Confidence Scale (ABC) | Change from Baseline (mean score at weeks 1, 2, 3, and 4) to Follow-Up (mean score at weeks 8, 12, 16, 20, 24, and 28)
  Self-report computerized survey (18 questions).
Patient Reported Outcomes Measurement Information System (PROMIS) | Change from Baseline (mean score at weeks 1, 2, 3, and 4) to Follow-Up (mean score at weeks 8, 12, 16, 20, 24, and 28)
  Self-report computerized questionnaire with 8-14 questions per domain. Includes Physical Function, Fatigue, and General Health subdomains.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Hafner, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Result] Hafner BJ, Askew RL. Physical performance and self-report outcomes associated with use of passive, adaptive, and active prosthetic knees in persons with unilateral, transfemoral amputation: Randomized crossover trial. J Rehabil Res Dev. 2015;52(6):677-700. doi: 10.1682/JRRD.2014.09.0210. PMID 26560243